CLINICAL TRIAL: NCT02726776
Title: Suspension Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A.10
Record Dates: First submitted 2016-03-15; First posted 2016-04-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Circulatory Collapse; Circulatory Failure; Syncope, Vasovagal, Neurally-Mediated; Orthostatic Hypotension
MeSH Terms: conditions — Shock; Syncope, Vasovagal; Hypotension, Orthostatic | interventions — Suspensions; Stair Climbing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suspension without prior climbing (Experimental): Free Suspension in a harness after baseline measurements and without prior climbing
  Interventions: Other: Suspension in a harness
- Suspension with prior climbing (Experimental): Free Suspension in a harness after baseline measurements and after climbing in moderate intensity for 10 minutes
  Interventions: Other: Suspension in a harness; Other: Climbing

INTERVENTIONS:
Other: Suspension in a harness
Other: Climbing
  Arms: Suspension with prior climbing

SUMMARY:
Suspension syndrome refers to a potentially life-threatening condition that can occur in unconscious persons after prolonged suspension in a harness. To date, our understanding of the pathophysiology and appropriate treatment is based primarily on case reports and expert opinion. The main pathophysiological hypothesis implicates blood pooling in the lower extremity and lack of return via muscle pumping. However, a recent French study could not support this hypothesis. Other mechanisms, such as a central vagal reflex may play a role in the pathophysiology of suspension syndrome. The aim of this study is to better understand the pathophysiological basis of suspension syndrome and to develop practical recommendations for prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-50 years
* ASA class 1
* Signed informed consent

Exclusion Criteria:

* Age <18 or >50 years
* ASA class >1
* Informed consent not signed

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Heart rate | Change from baseline (measurement at minute 0) -> suspension phase (minute 10, timepoint immediately before interruption of suspension phase [max 60 minutes]) -> minute 5 and minute 15 after suspension phase
Blood pressure | Change from baseline (measurement at minute 0) -> suspension phase (minute 10, timepoint immediately before interruption of suspension phase [max 60 minutes]) -> minute 5 and minute 15 after suspension phase

SECONDARY OUTCOMES:
Change in maximal Diameter of superficial femoral vein | Change from baseline (measurement at minute 0) -> suspension phase (minute 10, timepoint immediately before interruption of suspension phase [max 60 minutes]) -> minute 5 and minute 15 after suspension phase
  Ultrasound measurement of the Diameter of the superficial femoral vein in millimeters
Change in interbeat-interval | Change from baseline (measurement at minute 0) -> suspension phase (minute 10, timepoint immediately before interruption of suspension phase [max 60 minutes]) -> minute 5 and minute 15 after suspension phase
  electrocardiographic measurement of interbeat interval in milliseconds (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Paal, MD, MBA, Study Director — Barts Heart Centre, London; Hermann Brugger, MD, Study Director — Eurac, Institute of mountain emergency medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pasquier M, Yersin B, Vallotton L, Carron PN. Clinical update: suspension trauma. Wilderness Environ Med. 2011 Jun;22(2):167-71. doi: 10.1016/j.wem.2010.12.006. Epub 2010 Dec 23. PMID 21420883
- [Result] Lee C, Porter KM. Suspension trauma. Emerg Med J. 2007 Apr;24(4):237-8. doi: 10.1136/emj.2007.046391. PMID 17384373
- Available data/document: Study Protocol — https://cloud.scientificnet.org/index.php/s/7vKbCJ1vs0UOYNN — Unfortunately available only in German
- Available data/document: Informed Consent Form — https://cloud.scientificnet.org/index.php/s/9RXyWhRxEgUgbTd — Unfortunately available only in German or Italian